CLINICAL TRIAL: NCT04797273
Title: Internet-based Cognitive Behavior Therapy for Stress-related Disorders
Brief Title: Internet-based CBT vs. TAU for Stress-related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICBT vs TAU for Stress
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Adjustment Disorders; Exhaustion Disorder
Keywords: Internet-based treatment; Randomized controlled trial
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based cognitive behavior therapy (Experimental)
  Interventions: Behavioral: Internet-based cognitive behavior therapy
- Internet-based structured treatment-as-usual (Active Comparator)
  Interventions: Behavioral: Internet-based structured treatment-as-usual

INTERVENTIONS:
Behavioral: Internet-based cognitive behavior therapy — 12 week Internet-based cognitive behavior therapy, delivered via an online treatment platform. The treatment includes components such as exercises in conducting recuperating activities, methods to improve sleep, exposure, and behavioral activation. The treatment content is provided through written texts, images and audiofiles in the treatment platform. The participant has access to a therapist who provides support throughout the treatment via asynchronous text messages.
  Arms: Internet-based cognitive behavior therapy
Behavioral: Internet-based structured treatment-as-usual — This is a 12-week treatment, delivered via an online treatment platform. The treatment components in this treatment are designed to be similar to what is typically provided in primary care to these patients and includes information about stress and how different factors such as eating habits, physical exercise, and alcohol can contribute to stress problems. The treatment content is provided through written texts, images and audiofiles in the treatment platform. The participant has access to a therapist who provides support throughout the treatment via asynchronous text messages.
  Arms: Internet-based structured treatment-as-usual

SUMMARY:
Stress-related mental illness is common and one of the main causes of sick leave in Sweden. Cognitive behavior therapy (CBT) is a promising treatment, but access to treatment is low. In a previously conducted study, we found that internet-based CBT in comparison to a waitlist control group was effective in reducing symptoms of stress. The aim of the present study is to take the next step and compare Internet-based CBT for stress-related disorders to an active control condition.

DETAILED DESCRIPTION:
Non traumatic stress-related mental illness, in this study operationalized as adjustment disorder or exhaustion disorder, is highly prevalent in the general population and associated with high societal costs relating to productivity loss. Cognitive behavior therapy (CBT) is the most well-studied psychological treatment and has demonstrated promising effects in terms of symptom reduction. The overall evidence-base for CBT for these disorders is however fairly week and access to treatment is low. In a previously published randomized controlled trial we found that internet-based CBT can yield large effects on core symptoms of stress for these disorders. Delivering CBT via the internet has the large advantage of enabling increased accessibility as each therapist can have up to 80 patients in ongoing treatment. In the previously conducted trial we compared the treatment to a waitlist control and between-group comparisons of treatment effects were only done at post-treatment as the waitlist condition was crossed over to treatment after this time point. It is now therefore important to take the next step and investigate the effects of internet-based CBT in comparison to an active control condition. The primary aim of this study was to compare two internet-based treatments, CBT vs. structured treatment-as-usual, for adjustment disorder and exhaustion disorder.

ELIGIBILITY:
Inclusion Criteria:

* primary adjustment disorder or exhaustion disorder
* regular access to a computer and to the internet
* ability to read and write in swedish

Exclusion Criteria:

* substance abuse in the past 6 months
* lifetime psychosis or bipolar disorder
* suicide risk
* initiated or changed psychopharmacological treatment for depression or anxiety in the past month
* concurrent psychological treatment
* cognitive behavior therapy for stress-related symptoms in the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in PSS at post-treatment and follow-ups compared to baseline (scale range 0-40, higher score means more symptoms)

SECONDARY OUTCOMES:
Shirom-Melamed Burnout Questionnaire (SMBQ) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in SMBQ at post-treatment and follow-ups compared to baseline (scale range 1-7, higher score means more symptoms)
Montgomery-Åsberg Depression Rating Scale Self-report (MADRS-S) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in MADRS-S at post-treatment and follow-ups compared to baseline (scale range 0-54, higher score means more symptoms)
Insomnia Severity Index (ISI) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in ISI at post-treatment and follow-ups compared to baseline (scale range 0-28, higher score means more symptoms)
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in GAD-7 at post-treatment and follow-ups compared to baseline (scale range 0-21, higher score means more symptoms)
Sickness Questionnaire (SQ) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in SQ at post-treatment and follow-ups compared to baseline (scale range 0-30, higher score means more symptoms)
Self-rated Health (SRH) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in SRH at post-treatment and follow-ups compared to baseline (scale range 1-5, higher score means better self-rated health)
World Health Organization's Disability Assessment Scale (WHODAS 2.0) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in WHODAS at post-treatment and follow-ups compared to baseline (scale range 0-100, higher score means more functional disability)
EuroQol 5D (EQ5D 5L) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in EQ5D at post-treatment and follow-ups compared to baseline (The answers given in EQ-5D were combined to generate a utility score of health states ranging from 0 to 1, with 0 representing death and 1 representing full health) death and 1 representing full health
Trimbos and Institute Medical Technology Assessment of Costs Questionnaire for Psychiatry (TIC-P) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  The TIC-P enables estimation of costs by collecting information about participant resource utilization and costs related to production loss. Change in costs will be analysed at post-treatment and follow-ups compared to baseline.
Physical Health Questionnaire (PHQ-15) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Change in PHQ-15 at post-treatment and follow-ups compared to baseline (scale range 0-30, higher score means more symptoms)
Cognitive impairment | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Test-battery of cognitive tests measuring executive functions at post-treatment and follow-ups compared to baseline
Sick leave | 1 year prior to baseline up to 2 years after baseline.
  Sick leave data from the Microdata for Analysis of Social Security (MiDAS) registry. Analyzed as full-day equivalents.

OTHER OUTCOMES:
Karolinska Exhaustion Disorder Scale (KEDS) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Exploratory assessment of change at post-treatment and follow-ups compared to baseline (scale range 0-54, higher score means more symptoms)
Negative Events Questionnaire, 20-items (NEQ-20) | week 12 (Post-treatment)
  Post-treatment only report of negative events from treatment (scale range 0-80, higher score indicates more negative events)
Credibility scale (C-scale) | week 3
  week 3 only report of treatment credibility (scale range 0-50, higher score means higher credibility)
The Corona Virus Health Impact Survey -Short (CRISIS short) | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Exploratory analysis of the impact of the Corona virus on worry and life style. Change in sum score of items 1,2,3,4,5,8 and 9 will be analyzed. Scale range 0-24. Higher scores mean higher impact of Corona.
Subjective memory | Baseline, week 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Exploratory analysis of change in subjective memory at post-treatment and follow-ups compared to baseline (scale range 0-26, higher score means more subjective problems with memory)
Recovery Experience Questionnaire short version | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up, 2-year follow-up
  Will be analyzed as potential mediator of treatment change. 7 items, scored 0-4. Scale-range 0-28. Higher scores indicate more recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavsbergs Primary Care Center, Gustavsberg, Stockholm County, Sweden

REFERENCES:
- [Derived] Sennerstam V, Franke Foyen L, Kontio E, Svardman F, Lekander M, Lindsater E, Hedman-Lagerlof E. Internet-Delivered Treatment for Stress-Related Disorders: A Randomized Controlled Superiority Trial of Cognitive Behavioral Therapy versus General Health Promotion. Psychother Psychosom. 2025;94(4):273-288. doi: 10.1159/000546221. Epub 2025 May 7. PMID 40334656
- [Derived] Franke Foyen L, Sennerstam V, Kontio E, Lekander M, Hedman-Lagerlof E, Lindsater E. Objective cognitive functioning in patients with stress-related disorders: a cross-sectional study using remote digital cognitive testing. BMC Psychiatry. 2023 Aug 7;23(1):565. doi: 10.1186/s12888-023-05048-5. PMID 37550693